CLINICAL TRIAL: NCT05811949
Title: Effects of Dimethyl Fumarate on Cognitive Performances and Gray Matter and Thalamic Pathology in Multiple Sclerosis: a Correlation Study.
Brief Title: Effects of Dimethyl Fumarate on Cognitive Performance and Brain Abnormalities in Multiple Sclerosis.
Status: Completed | Type: Observational
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Sponsor
Other Study IDs: MSDMF_2020
Record Dates: First submitted 2023-03-17; First posted 2023-04-13 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Dimethyl Fumarate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- RRMS patients with de novo DMF treatment: RRMS patients with de novo treatment who start DMF.
  Interventions: Drug: Dimethyl Fumarate 240 MG [Tecfidera]
- RRMS patients switching to DMF.: RRMS patients who switch from first-line DMT treatment (interferon, glatiramer acetate, teriflunomide) to treatment with DMF.
  Interventions: Drug: Dimethyl Fumarate 240 MG [Tecfidera]

INTERVENTIONS:
Drug: Dimethyl Fumarate 240 MG [Tecfidera] — DMF is admnistered to RRMS patients who are candidates for treatment according to clinical practice at a dosage of 120 mg twice daily, increased to 240 mg twice daily after 7 days.

SUMMARY:
The goal of this observational study is to evaluate the slowing/reduction of cognitive dysfunction progression and to evaluate grey matter (GM) and thalamus structural changes in Relapsing-Remitting Multiple Sclerosis (RRMS) patients after 12 months of treatment with Dimethyl Fumarate (DMF).

The main questions it aims to answer are:

* Can DMF slow or reduce the progression of cognitive dysfunction in RRMS patients?
* Can DMF slow the reduction of brain volume in RRMS patients?

At baseline visit, RRMS patients undergo extensive neurological examination in which their disability is evaluated by using Expanded Disability Status Scale (EDSS). The efficacy assessments of this study are:

1. The Brief Repeatable Neuropsychological Battery (BRB);
2. Executive functions: Delis-Kaplan Function System (DKEFS) scale - Sorting Test.

All RRMS patients undergo MRI: conventional MRI measures (T2-, T1-enhancing and T1-hypointense lesions), global brain atrophy, regional brain atrophy and Diffusion Tensor Imaging (DTI) (GM and thalamus) examinations.

Six and 12 months after the baseline visit, the RRMS patients in treatment with DMF undergo the BRB, DKEFS and MRI/DTI study and neurological evaluation (EDSS).

DETAILED DESCRIPTION:
Dimethyl fumarate (DMF) is an oral disease-modifying therapy (DMT) approved for management of Relapsing-Remitting Multiple Sclerosis (RRMS) patients. Clinical trials have shown that DMF has a significant beneficial impact on relapse rate, disability accrual and the number of new lesions along with their volumes. In addition, a neuroprotective role of DMF has been suggested to occur on both the gray matter (GM) and thalamus. However, there are no correlation data in the literature between the effects of DMF on cognitive performance and those on the GM, with a focus on thalamic pathology in MS patients.

The primary objectives of this study are:

i) to evaluate the slowing/reduction of cognitive dysfunction progression in RRMS patients after 12 months of treatment with DMF; ii) to evaluate the effects of DMF on Magnetic Resonance Imaging (MRI) parameters in GM and thalamus.

The secondary objective is to evaluate how the effects on cognitive dysfunction progression are associated to the effect of slowing the brain volume reduction at MRI (antiatrophic effect) and to change of Diffusion Tensor Imaging (DTI) parameters that DMT might have in RRMS patients, in the GM and thalamus.

The tertiary objective is to assess whether differences exist between patients with RRMS de novo to DMF treatment and patients switching from first-line DMT to DMF.

After signing informed consent, demographics, medical history and current therapies are collected for each RRMS patient enrolled. RRMS patients undergo extensive neurological examination in which their disability is evaluated by using EDSS. The efficacy assessments of this study are:

1. The Brief Repeatable Neuropsychological Battery (BRB)
2. Executive functions: Delis-Kaplan Function System (DKEFS) scale - Sorting Test.

All MS patients undergo MRI: conventional MRI measures (T2-, T1-enhancing and T1-hypointense lesions), global brain atrophy, regional brain atrophy and DTI (GM and thalamus) examinations.

Six and 12 months after the baseline visit, the RRMS patients in treatment with DMF undergo the BRB, DKEFS and MRI/DTI study and neurological evaluation (EDSS).

ELIGIBILITY:
Inclusion Criteria:

* Patients must voluntarily give written informed consent. Patients must read and fully understand the Informed Consent Form (ICF);
* Patient diagnosed with MS according to McDonald criteria;
* Adult patients, males or female patients ≥ 18 years old;
* Relapsing disease course;
* Expanded Disability Status Scale (EDSS) ≤5.5;
* Patients who initiate treatment with DMF 240 mg twice daily according prescribing criteria.

Exclusion Criteria:

* Diagnosis of non-relapsing MS;
* Use of experimental drug or investigational procedure during the study period;
* Pregnancy;
* Severe hepatic impairment;
* Relapse or corticosteroid use within 30 days prior to baseline MRI scan;
* Previous use of alemtuzumab, cladribine, rituximab, or mitoxantrone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is conducted in 52 patients: twenty-six de novo MS patients who start DMF treatment and 26 patients who switch from first-line DMT treatment (interferon, glatiramer acetate, teriflunomide) to treatment with DMF are matched for age and gender. Sample size calculation considers a significance level of 5% and a power of 80% to detect a difference of 0.22 with a standard deviation of 0.5, assuming a patients' loss of 20-30%.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Change in subjects' cognitive performance | Month 0 Baseline to Month 6 Follow-up
  Change from baseline in Selective Reminding Test - Long-Term Storage (SRT-LTS) Raw Score of Brief Repeatable Battery (BRB) at 6 months. This is one of the five tests of BRB for episodic memory (verbal learning and delayed recall). A word recalled on two consecutive trials is considered to have entered long-term storage (LTS) on the first of these trials and scored as LTS on all following trials. The total score ranged from 0 to 72. Higher values represent a better outcome.
Change in subjects' cognitive performance | Month 0 Baseline to Month 6 Follow-up
  Change from baseline in Selective Reminding Test - Consistent Long Term Retrieval (SRT-CLTR) Raw Score of Brief Repeatable Battery (BRB) at 6 months. This is one of the five tests of BRB for episodic memory (verbal learning and delayed recall). A word recalled on two consecutive trials is considered to have entered long-term storage (LTS) on the first of these trials and scored as LTS on all following trials. The total of the words in LTS of all six trials is then summed. If a word in LTS is consistently recalled on all subsequent trials, it is then scored as Consistent Long Term Retrieval (CLTR). The total of the words in CLTR of all six trials is summed. The total score ranged from 0 to 72. Higher values represent a better outcome.
Change in subjects' cognitive performance | Month 0 Baseline to Month 6 Follow-up
  Change from baseline in Spatial Recall Test (SPART) Raw Score of Brief Repeatable Battery (BRB) at 6 months. The spatial recall test assesses visuospatial learning and delayed recall. The total score ranged from 0 to 30. Higher values represent a better outcome.
Change in subjects' cognitive performance | Month 0 Baseline to Month 6 Follow-up
  Change from baseline in Symbol Digit Modalities Test (SDMT) Raw Score of Brief Repeatable Battery (BRB) at 6 months. Symbol Digit Modality Test (SDMT) for sustained attention and information processing speed. The score is the number of correct answers in 90 seconds. The total score ranged from 0 to 110. Higher values represent a better outcome.
Change in subjects' cognitive performance | Month 0 Baseline to Month 6 Follow-up
  Change from baseline in Paced Auditory Serial Addition Test - 3 Seconds (PASAT 3) Raw Score of Brief Repeatable Battery (BRB) at 6 months. Paced Auditory Serial Addition Test (PASAT) for working memory (and sustained attention and information processing speed). The total score ranged from 0 to 60. Higher values represent a better outcome.
Change in subjects' cognitive performance | Month 0 Baseline to Month 6 Follow-up
  Change from baseline in Paced Auditory Serial Addition Test - 2 (PASAT 2) Raw Score of Brief Repeatable Battery (BRB) at 6 months. Paced Auditory Serial Addition Test (PASAT) for working memory (and sustained attention and information processing speed). The total score ranged from 0 to 60. Higher values represent a better outcome.
Change in subjects' cognitive performance | Month 0 Baseline to Month 6 Follow-up
  Change from baseline in Selective Reminding Test - Delayed Recall (SRT-D) Raw Score of Brief Repeatable Battery (BRB) at 6 months. The tests SRT (Selective Reminding Test) for episodic memory (verbal learning and delayed recall).The total score ranged from 0 to 12. Higher values represent a better outcome.
Change in subjects' cognitive performance | Month 0 Baseline to Month 6 Follow-up
  Change from baseline in Spatial Recall Test - Delayed Recall (SPART-D) of Brief Repeatable Battery (BRB) at 6 months. Spatial Recall Test (SPART) for visuospatial learning and delayed recall. Spatial Recall Test (10/36): The spatial recall test assesses visuospatial learning and delayed recall (10/36-D). The total score ranged from 0 to 10. Higher values represent a better outcome.
Change in subjects' cognitive performance | Month 0 Baseline to Month 6 Follow-up
  Change from baseline in Word List Generation (WLG) of Brief Repeatable Battery (BRB) at 6 months. Word List Generation (COWAT/WLG): The COWAT assesses verbal fluency on semantic stimulus by asking the patient to produce as many words as possible belonging to a semantic category. No maximum range is available. Higher values represent a better outcome. The score is the number of correct words. The more words the patient pronounces, the better it is. We can imagine that the minimum value might be zero words, but it is not a score scale.
Change in subjects' cognitive performance | Month 0 Baseline to Month 12 Follow-up
  Change from baseline in Selective Reminding Test - Long-Term Storage (SRT-LTS) Raw Score of Brief Repeatable Battery (BRB) at 12 months. One of the five tests of BRB is SRT (Selective Reminding Test) for episodic memory (verbal learning and delayed recall). A word recalled on two consecutive trials is considered to have entered long-term storage (LTS) on the first of these trials and scored as LTS on all following trials. The total score ranged from 0 to 72. Higher values represent a better outcome.
Change in subjects' cognitive performance | Month 0 Baseline to Month 12 Follow-up
  Change from baseline in Selective Reminding Test - Consistent Long Term Retrieval (SRT-CLTR) Raw Score of Brief Repeatable Battery (BRB) at 12 months. One of the five tests of BRB is SRT (Selective Reminding Test) for episodic memory (verbal learning and delayed recall). A word recalled on two consecutive trials is considered to have entered long-term storage (LTS) on the first of these trials and scored as LTS on all following trials. The total of the words in LTS of all six trials is then summed. If a word in LTS is consistently recalled on all subsequent trials, it is then scored as Consistent Long Term Retrieval (CLTR). The total of the words in CLTR of all six trials is summed. The total score ranged from 0 to 72. Higher values represent a better outcome.
Change in subjects' cognitive performance | Month 0 Baseline to Month 12 Follow-up
  Change from baseline in Spatial Recall Test (SPART) Raw Score of Brief Repeatable Battery (BRB) at 12 months. The spatial recall test assesses visuospatial learning and delayed recall. The total score ranged from 0 to 30. Higher values represent a better outcome.
Change in subjects' cognitive performance | Month 0 Baseline to Month 12 Follow-up
  Change from baseline in Symbol Digit Modalities Test (SDMT) Raw Score of Brief Repeatable Battery (BRB) at 12 months. Symbol Digit Modality Test (SDMT) for sustained attention and information processing speed. The score is the number of correct answers in 90 seconds. The total score ranged from 0 to 110. Higher values represent a better outcome
Change in subjects' cognitive performance | Month 0 Baseline to Month 12 Follow-up
  Change from baseline in Paced Auditory Serial Addition Test - 3 Seconds (PASAT 3) Raw Score of Brief Repeatable Battery (BRB) at 12 months. Paced Auditory Serial Addition Test (PASAT) for working memory (and sustained attention and information processing speed). The total score ranged from 0 to 60. Higher values represent a better outcome.
Change in subjects' cognitive performance | Month 0 Baseline to Month 12 Follow-up
  Change from baseline in Paced Auditory Serial Addition Test - 2 (PASAT 2) Raw Score of Brief Repeatable Battery (BRB) at 12 months. +Paced Auditory Serial Addition Test (PASAT) for working memory (and sustained attention and information processing speed). The total score ranged from 0 to 60. Higher values represent a better outcome.
Change in subjects' cognitive performance | Month 0 Baseline to Month 12 Follow-up
  Change from baseline in Selective Reminding Test - Delayed Recall (SRT-D) Raw Score of Brief Repeatable Battery (BRB) at 12 months. The tests SRT (Selective Reminding Test) for episodic memory (verbal learning and delayed recall).The total score ranged from 0 to 12. Higher values represent a better outcome.
Change in subjects' cognitive performance | Month 0 Baseline to Month 12 Follow-up
  Change from baseline in Spatial Recall Test - Delayed Recall (SPART-D) of Brief Repeatable Battery (BRB) at 12 months. Spatial Recall Test (SPART) for visuospatial learning and delayed recall.Spatial Recall Test (10/36): The spatial recall test assesses visuospatial learning and delayed recall (10/36-D). The total score ranged from 0 to 10. Higher values represent a better outcome.
Change in subjects' cognitive performance | Month 0 Baseline to Month 12 Follow-up
  Change from baseline in Word List Generation (WLG) of Brief Repeatable Battery (BRB) at 12 months. Word List Generation (COWAT/WLG): The COWAT assesses verbal fluency on semantic stimulus by asking the patient to produce as many words as possible belonging to a semantic category. No maximum range is available. Higher values represent a better outcome. The score is the number of correct words. The more words the patient pronounces, the better it is. We can imagine that the minimum value might be zero words, but it is not a score scale.
Change in subjects' cognitive performance | Month 0 Baseline to Month 6 Follow-up
  Change from baseline in Delis-Kaplan Executive Function System (DKEFS) Condition 1: Free Sorting, Confirmed Correct Sort - Card Set 1+2 at 6 months. The standard form consists of the practice card set, card set 1 and card set 2. The alternate form consists of the same practice card set, card set 3 and card set 4. The DKFES test consisted of two testing procedures: free sorting and sort recognition. In free sorting, six scores are obtained: Confirmed Correct sorts for card sets 1 and 2 (or 3 and 4 for version B), sum of confirmed Correct Sorts. In sort recognition, a description score for card set 1 and 2 (or 3 and 4 for version B) is obtained, as well as the sum of description scores of both sets. The total score ranges from 0 to 16. Higher values represent a better outcome.
Change in subjects' cognitive performance | Month 0 Baseline to Month 6 Follow-up
  Change from baseline in DKEFS Condition 1: Free Sorting, Free Sorting, Description Score, Card Set 1+2 at 6 months. The standard form consists of the practice card set, card set 1 and card set 2. The alternate form consists of the same practice card set, card set 3 and card set 4. In free sorting, six scores were obtained: Confirmed Correct sorts for card sets 1 and 2 (or 3 and 4 for version B), sum of confirmed Correct Sorts, Free Sorting Description score for card set 1 and 2 (or 3 and 4 for version B) and sum of Free Sorting Description scores. In sort recognition, a description score for card set 1 and 2 (or 3 and 4 for version B) was obtained, as well as the sum of description scores of both sets. The total score ranged from 0 to 64. Higher values represent a better outcome.
Change in subjects' cognitive performance | Month 0 Baseline to Month 6 Follow-up
  Change from baseline in DKEFS Condition 2: Sort Recognition, Sort Recognition Description Score- Card Set 1+22 at 6 months. The standard form consists of the practice card set, card set 1 and card set 2. The alternate form consists of the same practice card set, card set 3 and card set 4. Free sorting and sort recognition. In free sorting, six scores were obtained: Confirmed Correct sorts for card sets 1 and 2 (or 3 and 4 for version B), sum of confirmed Correct Sorts, Free Sorting Description score for card set 1 and 2 (or 3 and 4 for version B) and sum of Free Sorting Description scores. The total score ranged from 0 to 64. Higher values represent a better outcome.
Change in subjects' cognitive performance | Month 0 Baseline to Month 12 Follow-up
  Change from baseline in Delis-Kaplan Executive Function System (DKEFS) Condition 1: Free Sorting, Confirmed Correct Sort - Card Set 1+2 at 12 months. The standard form consists of the practice card set, card set 1 and card set 2. The alternate form consists of the same practice card set, card set 3 and card set 4. The DKFES test consisted of two testing procedures: free sorting and sort recognition. In free sorting, six scores are obtained: Confirmed Correct sorts for card sets 1 and 2 (or 3 and 4 for version B), sum of confirmed Correct Sorts. In sort recognition, a description score for card set 1 and 2 (or 3 and 4 for version B) is obtained, as well as the sum of description scores of both sets. The total score ranges from 0 to 16. Higher values represent a better outcome.
Change in subjects' cognitive performance | Month 0 Baseline to Month 12 Follow-up
  Change from baseline in DKEFS Condition 1: Free Sorting, Free Sorting, Description Score, Card Set 1+2 at 12 months. The standard form consists of the practice card set, card set 1 and card set 2. The alternate form consists of the same practice card set, card set 3 and card set 4. In free sorting, six scores were obtained: Confirmed Correct sorts for card sets 1 and 2 (or 3 and 4 for version B), sum of confirmed Correct Sorts, Free Sorting Description score for card set 1 and 2 (or 3 and 4 for version B) and sum of Free Sorting Description scores. In sort recognition, a description score for card set 1 and 2 (or 3 and 4 for version B) was obtained, as well as the sum of description scores of both sets. The total score ranged from 0 to 64. Higher values represent a better outcome.
Change in subjects' cognitive performance | Month 0 Baseline to Month 12 Follow-up
  Change from baseline in DKEFS Condition 2: Sort Recognition, Sort Recognition Description Score - Card Set 1+22 at 12 months. The standard form consists of the practice card set, card set 1 and card set 2. The alternate form consists of the same practice card set, card set 3 and card set 4. Free sorting and sort recognition. In free sorting, six scores were obtained: Confirmed Correct sorts for card sets 1 and 2 (or 3 and 4 for version B), sum of confirmed Correct Sorts, Free Sorting Description score for card set 1 and 2 (or 3 and 4 for version B) and sum of Free Sorting Description scores. The total score ranged from 0 to 64. Higher values represent a better outcome.
Changes brain MRI parameters | Month 0 Baseline to Month 6 Follow-up
  Change from baseline GM and thalamus volume at 6 months.
Changes brain MRI parameters | Month 0 Baseline to Month 12 Follow-up
  Change from baseline GM and thalamus volume at 12 months.
Changes brain MRI parameters | Month 0 Baseline to Month 6 Follow-up
  Change from baseline DTI measures in the GM and thalamus at 6 months.
Changes brain MRI parameters | Month 0 Baseline to Month 12 Follow-up
  Change from baseline DTI measures in the GM and thalamus at 12 months.

SECONDARY OUTCOMES:
Correlation between scores of cognitive battery and brain MRI parameters | Baseline and 6 and 12 months after.
  Correlation data between each test of cognitive battery, in terms of mean changes in total score observed at endpoint vs. baseline, and brain volume reduction and DTI parameters (in GM and thalamus), as mean change after 12 months of treatment.

OTHER OUTCOMES:
Difference between the two cohorts | Baseline and 6 and 12 months after.
  Difference between the two cohorts in terms of mean changes in total score of BRB and DKEFS scale and in terms of mean changes in brain volume and DTI parameters (in GM and thalamus).

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Centro Neurolesi "Bonino-Pulejo", Messina, Italy

IPD SHARING:
Plan to Share IPD: Undecided